CLINICAL TRIAL: NCT02100085
Title: A Single Center, Phase I Study to Follow-up on the Change of Immunogenicity and Lesion Condition in Subjects Who Have Completed the Phase I GX-188E Trial (Protocol no. GX-188E-SN)
Brief Title: Safety and Efficacy of GX-188E DNA Therapeutic Vaccine Administered by Electroporation After Observation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GX-188E-FU
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Cervical Intraepithelial Neoplasia 3
Keywords: Phase 1 follow up; Cervical Intraepithelial Neoplasia; Adult; Safety; Efficacy
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — GX-188 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and PBMC (peripheral blood mononeuclear cells)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational group: Subjects in the period less than 48 weeks after the final administration of GX-188E
  Interventions: Biological: GX-188E

INTERVENTIONS:
Biological: GX-188E — In phase I study, 9 patients were assigned to three dose groups (1mg, 2mg and 4mg) and were administered three times with GX-188E by electroporation during an entire period of study. After the final administration, the follow-up will be conducted to investigate safety and efficacy aspects.
  Other Names: GX-188E administerd by eletrophoration

SUMMARY:
This study is to follow up on the change of immune response by measuring HPV type 16/18 E6 and E7 specific T cell response and lesion condition in subjects who have administered in DNA-based therapeutic vaccine.

DETAILED DESCRIPTION:
This is a follow-up study to investigate the change of immunogenicity and lesion condition in subjects with cervical intraepithelial neoplasia (CIN) 3 who have enrolled and completed GX-188E phase I study.

Subjects will make visits at week 48 (V1) to week 228 (V8) every 6 months after the final administration of GX-188E.

The endpoints are to evaluate the change of immune response, involved lesion and infection status compared to that of the final visit in phase I study.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 20 and 50 (inclusive)
* The subjects who have visited within 48 weeks after final injection of GX-188E
* Those who voluntarily signed informed consent form

Exclusion Criteria:

* Prior participation in any clinical trial within 30 days prior to the visit 1
* Any other ineligible condition at the discretion of the investigator that would be ineligible to participate the study

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subjects who have completed the DNA vaccine administration of each dosage (1, 2 and 4 mg).
  The subjects in the period less than 48 weeks after the final administration of GX-188E
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The change of the immune response compared to that of the final visit in phase I study | at week 0 to 180 every 6 months
  It would be determined by evaluating HPV type 16/18 E6 and E7 specific T cell response (IFN-γ ELISPOT assay) using PBMC obtained at week 0 to 180 visit every 6 months.

SECONDARY OUTCOMES:
The change of the involved lesion and HPV infection status | at week 0 to 180 every 6 months
  The changes of histological test, cytological test and HPV infection status would be compared to that of the last visit in phase I study
Safety profile | at week 0 to 180 every 6 months
  Safety profile would be examined by vital signs, physical examination, clinical laboratory tests etc

CONTACTS AND LOCATIONS:
Overall Officials: Tae Jin Kim, M.D., Principal Investigator — Cheil General Hospital & Women's Healthcare Center
Locations (1):
- Cheil General Hospital & Women's Healthcare Center, Seoul, Korea, South Korea